CLINICAL TRIAL: NCT04799080
Title: Investigation of the Effect of Chemotherapy-induced Peripheral Neuropathy (CIPN) on Sensory and Motor Function in Patients With Cancer
Brief Title: Chemotherapy-induced Peripheral Neuropathy (CIPN) on Motor and Sensory Function
Status: Completed | Type: Observational
Sponsor: Izmir Bakircay University (Other)
Responsible Party: Principal Investigator, Alper Tuğral, PT, MSc, Izmir Bakircay University
Other Study IDs: BakircayU/D208
Record Dates: First submitted 2021-03-11; First posted 2021-03-16 (Actual); Last update posted 2024-04-01 (Actual); Status verified 2024-03

CONDITIONS: Cancer; Chemotherapy-induced Peripheral Neuropathy; Chemotherapeutic Toxicity; Breast Cancer; Breast Neoplasms; Colon Neoplasm; Colo-rectal Cancer
Keywords: Chemotherapy-induced Peripheral Neuropathy; Hand Grip; Cutaneous; Quality of Life
MeSH Terms: conditions — Neoplasms; Breast Neoplasms; Colonic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
As cancer survival rates have been increased due to technological developments and early detection strategies, there has been been a growing need to assess the effect of long-term complications and adverse effects upon patients' functionality and quality of life. Chemotherapy, which is accepted to be the body of systemic adjuvant therapy is attributed to long-term survival, yet some side effects such as sarcopenia, loss of muscle strength and functional capacity, fatigue, and sensory disturbances due to the neurotoxic effects have been well known. Chemotherapy-induced peripheral neuropathy (CIPN) is a condition that is characterized by main loss of cutaneous sensation especially in the distal part of the extremities. CIPN affects approximately 30-40% of patients with cancer undergoing chemotherapy. Loss of sensation in distal sides of upper and lower extremities may cause not only deterioration of fine hand skills but also loss of balance and thereby one's mobility and independence are detrimentally affected. Thus, this study is aimed to assess CIPN in patients with cancer undergoing chemotherapy in a longitudinal design by assessing the cutaneous function of the sensory nerves and related effect of motor function.

DETAILED DESCRIPTION:
Chemotherapy-induced peripheral neuropathy (CIPN) which affects over 30-40% of patients with cancer undergoing chemotherapy cause cutaneous loss of sensation. A specific and selective function carries great importance not only in daily life but also in task-specific complex movements. Since the long-term survival of cancer is increased, back to work is quite important in both one's participation in community life and financial issues. Irrespective of age or other socio-clinical and socio-demographic characteristics, patients may be affected detrimentally after systemic adjuvant chemotherapy implementation in the perspective of sensory and motor aspects. Thus, this study is aimed to assess cutaneous sensory and motor function in patients with cancer undergoing chemotherapy in a longitudinal design.

Study Setting:

This research was planned as an observational-cross sectional cohort study within a longitudinal design. Patients diagnosed with cancer and applied to medical oncology unit in Izmir Bakircay University Çiğli State and Training Hospital for systemic adjuvant chemotherapy will be assessed in three different time points set as following: Time 1: before chemotherapy application, Time 2: interim time point (approx.8 weeks later) and Time 3: post-chemotherapy time point (12-20 weeks later after initial assessment). The main outcome measures were set as handgrip strength and Minnesota Rate of Manipulation Test (MRMT) for motor function while Semmens-Weinstein Monofilament Test (SWMT) for sensory evaluation. Secondarily, patients' quality of life and fatigue will be assessed with European Organization of Research and Treatment of Cancer (EORTC) specific scales such as QLQ-C30 for general quality of life and QLQ-FA12 for fatigue.

Hand Grip Strength:

Hand-Grip Strength Handgrip strength will be assessed with Lafayette Professional Hand Dynamometer, Model 5030L1, LaFayette Instruments, NY, USA). The standard position which can be achieved by 90-degree elbow flexion, shoulder abducted, and hand mid-prone positioned; 90-degree shoulder abduction and 90-degree shoulder abduction positions will be used to assess hang-grip strength. Three measurements will be requested and the maximum value of them will be recorded.

MRMT:

The Minnesota Rate of Manipulation test (MRMT, LaFayatte Instruments, NY, USA) will be used to assess the fine hand skills of patients who undergo chemotherapy. There are five other sub-tests to evaluate hand function such as one or two hands turning, displacing, etc. However, since CIPN might affect both hands, we chose to use two hands turning and placing the test.

Briefly, 60 wooden circle-shaped discs are placed on the pegboard. (15 discs x 4 row). Patients are requested to stand in front of the pegboard. Each patient will be informed about the test as following: "Start with the top-right corner of the board. Hold the disc and turn with your right hand, give it to your left then place it again. Continue this until reaching the top left corner. In the second row, you will start to top left corner, hold the disc and turn with your left hand, give it to your right and place it again". Patients also will be informed about doing this as best and fast they can while avoiding exaggerated movements of the trunk. Each patient will be tested for two trials, the third one will be the main test in which time will be calculated via chronometer.

Scales and Forms:

There will be scales and form which are required to fill out by participants. The following list of scales will be filled with participants themselves.

The European Organization for Research and Treatment of Cancer Quality of Life Questionnaire (EORTC-QLQ-C30) is the most frequently used cancer-specific health-related questionnaire. It consists of 28 items and each is scored "1: None" through "4: A lot" according to the 4-based Likert Scoring System. Besides, Item 29 and 30 are scored "1" through "7" in which are asked about health and quality of life through the last week. The higher scores indicate the worst quality of life or vice versa.

EORTC-QLQ-BR23 is the sub-module of the C30 questionnaire which consists of a total of 23 items. Scoring and interpretation of the questionnaire total score are the same as with the C30 questionnaire. Patients diagnosed with breast cancer and who volunteered to participate in this study are also requested to fill out this health-related quality of life patient-reported outcome scale. While C30 is requested to fill out for all patients.

Functional Assessment of Cancer Therapy (FACT-B+) The Functional Assessment of Cancer Therapy- Breast (FACT-B) consists of 37 items. To assess the health-related specific quality of life of patients with breast cancer, each item is scored "0: None" through "4: A Lot". Emotional, Functional, Physical, Social, and Family and Other Concerns are the main sub-domains that directly assess the related quality of life. Higher scores indicate worst, while lower scores indicate the best.

Purpose of This Research:

1. To evaluate the effect of chemotherapy-induced peripheral neuropathy (CIPN) on the motor and sensory function
2. To compare results of functional capacity, motor and sensory function between pre-chemotherapy and post-chemotherapy

The hypothesis of this study:

H0: There is no difference in hand and plantar cutaneous sensory function between pre-chemotherapy and post-chemotherapy periods H1-1: Cutaneous function of both sides of the hand and plantar skin tissue is decreased due to chemotherapy.

H2-1: Functional capacity and quality of life are decreased due to chemotherapy compared to the baseline values.

H3-1: Handgrip strength and Hand dexterity test results are worsened due to chemotherapy compared to the baseline values.

Power Analysis:

A priori power analysis was performed via the G*Power 3.1.9 program. Since there will be repeated measures along with three different time points, a power analysis was performed according to the within-group factors design in repeated measures analysis of variance test. Middle effect size according to the partial eta squared was set at 0.03 then general effect size was calculated as 0.17. In 95% Confidence Interval and 80% power, setting non-sphericity correction as default and correlation among repeated measures was set as 0.5. It was found that a total of 54 participants are needed to achieve these results, however, in case of a 10% potential drop-out rate and possible violation of sphericity, it is planned to include a total of 72 patients in this study.

ELIGIBILITY:
Inclusion Criteria:

* Being a Volunteer to participate this study
* Having diagnosed with Cancer
* Having available to be implemented to adjuvant systemic chemotherapy application

Exclusion Criteria:

* Prior diagnosed with diabetic polyneuropathy
* Neo-adjuvant chemotherapy
* Having scar tissue in the palmar and/or plantar side(s) of the skin might affect the sensory evaluation
* Having Multiple Sclerosis or other neurological diseases which might affect neural conductivity disturbances and/or sensory loss

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with cancer especially with colon, colorectal, and breast who will undergo a systemic adjuvant chemotherapy implementation.
Sampling Method: Non-Probability Sample
Enrollment: 72 (Actual)
Dates: Start 2021-03-06 (Actual); Primary Completion 2022-03-15 (Actual); Study Completion 2022-05-15 (Actual)

PRIMARY OUTCOMES:
Hand Grip Strength | 6 weeks
  Motor Function Asssesment via Hand-Grip Strength
Minnesota Rate of Manipulation Test | 6 weeks
  Functional Assessment of Hands
Semmens Weinstein Monofilament Test (SWMT) | 6 weeks
  Evaluation of Cutaneous Sensory Function

SECONDARY OUTCOMES:
The European Organization for Research and Treatment of Cancer Quality of Life Questionnaire (EORTC-QLQ-C30) | 6 weeks
  Quality of Life Questionnaire
Functional Assessment of Cancer Therapy-Breast (FACT-B+) | 6 weeks
  Health Related Quality of Life Assessment

CONTACTS AND LOCATIONS:
Overall Officials: Murat Akyol, MD, Principal Investigator — Bakircay University Faculty of Medicine Department of Internal Medicine, Medical Oncology unit; Zeynep Arıbaş, PT, Principal Investigator — Bakircay University Faculty of Health Sciences Department of Physical Therapy and Rehabilitation; Alper Tuğral, PT, MSc, Principal Investigator — Bakircay University Faculty of Health Sciences Department of Physical Therapy and Rehabilitation; Yeşim Bakar, PT, Prof, Principal Investigator — Bakircay University Faculty of Health Sciences Department of Physical Therapy and Rehabilitation
Locations (1):
- Bakircay University Çiğli State and Training Hospital, Department of Medical Oncology, Izmir, Çiğli, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Staff NP, Grisold A, Grisold W, Windebank AJ. Chemotherapy-induced peripheral neuropathy: A current review. Ann Neurol. 2017 Jun;81(6):772-781. doi: 10.1002/ana.24951. Epub 2017 Jun 5. PMID 28486769
- [Background] Seretny M, Currie GL, Sena ES, Ramnarine S, Grant R, MacLeod MR, Colvin LA, Fallon M. Incidence, prevalence, and predictors of chemotherapy-induced peripheral neuropathy: A systematic review and meta-analysis. Pain. 2014 Dec;155(12):2461-2470. doi: 10.1016/j.pain.2014.09.020. Epub 2014 Sep 23. PMID 25261162
- [Background] Quasthoff S, Hartung HP. Chemotherapy-induced peripheral neuropathy. J Neurol. 2002 Jan;249(1):9-17. doi: 10.1007/pl00007853. PMID 11954874
- [Derived] Tugral A, Aribas Z, Akyol M, Bakar Y. Assessment of sensorimotor and strength related function of breast cancer patients during systemic drug therapy: a prospective observational study. BMC Cancer. 2023 Oct 14;23(1):981. doi: 10.1186/s12885-023-11494-x. PMID 37838686